CLINICAL TRIAL: NCT03008616
Title: A Phase 2b/3a, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of the Efficacy and Safety of AMAG-423, a Digoxin Immune Fab, in Antepartum Subjects With Severe Preeclampsia
Brief Title: Study of the Efficacy and Safety of AMAG-423 (Digoxin Immune Fab) in Antepartum Subjects With Severe Preeclampsia
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Following a recommendation from the Data and Safety Monitoring Board (DSMB), the study was stopped early for futility. There were no safety concerns raised.
Sponsor: AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMAG-423-201
Record Dates: First submitted 2016-12-20; First posted 2017-01-02 (Estimated); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Severe Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — digoxin antibodies Fab fragments

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AMAG-423 (digoxin immune fab) (Active Comparator): AMAG-423 (digoxin immune fab) 3.2 mg/kg, 30 minute IV infusion, every 6 hours x 4 days
  Interventions: Biological: AMAG-423 (digoxin immune fab)
- Placebo (Placebo Comparator): Normal saline, 30 minute IV infusion, every 6 hours x 4 days
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: AMAG-423 (digoxin immune fab) — AMAG-423 (digoxin immune fab) 3.2 mg/kg, 30 minute IV infusion, every 6 hours x 4 days
  Other Names: DigiFab
  Arms: AMAG-423 (digoxin immune fab)
Other: Placebo — Normal saline, 30 minute IV infusion, every 6 hours x 4 days
  Arms: Placebo

SUMMARY:
This study evaluates the use of AMAG-423 (Digoxin Immune Fab) in addition to expectant management in the treatment of severe preeclampsia as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Fetal gestational age 23 0/7 to 31 6/7 weeks
* Treated with expectant management
* Meets modified ACOG criteria for severe preeclampsia
* Willing and able to provide written, informed consent

Exclusion Criteria:

* Decision to deliver within 24 hours has been made
* Weight > 150 kg
* Eclampsia
* Significant antecedent obstetrical problems
* Clinically significant fetal anomaly or chromosomal abnormalities
* Chronic renal disease
* Active hepatic disease, antiphospholipid antibody syndrome, or lupus
* Unstable medical or psychiatric disorder
* Need for use of digitalis like products
* History of anaphylactic allergic reactions
* Prior use of antibodies/fab fragments from sheep
* Serum creatinine ≥ 2.0 mg/dL
* Platelet count < 50,000
* Pulmonary edema
* Estimated fetal weight < 5th percentile

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2020-08-13 (Actual); Study Completion 2020-08-13 (Actual)

PRIMARY OUTCOMES:
Proportion of infants who have severe IVH, NEC, or death by 36 weeks corrected gestational age | 36 weeks corrected gestational age
  Proportion of infants who have severe IVH, NEC, or death by 36 weeks corrected gestational age

SECONDARY OUTCOMES:
Change from baseline in serum creatinine | From treatment initiation to 24 hours post first dose
  Maternal change from baseline in serum creatinine to 24 hours post first dose
Incidence of pulmonary edema | From treatment initiation until completion of treatment phase (up to 4 days)
  Maternal incidence of pulmonary edema during the treatment period
Proportion of mothers with modified early obstetric warning score >= 3 at 24 hours post first dose | 24 hours post first dose
  Proportion of mothers with modified early obstetric warning score >= 3 at 24 hours post final dose
Delivery latency | From treatment initiation until delivery
  Time from start of treatment until delivery
Anti-hypertensive use during treatment | From treatment initiation until completion of treatment phase (up to 4 days)
  Use of or change in anti-hypertensive use during the treatment period

CONTACTS AND LOCATIONS:
Locations (18):
- United States (16):
  - University of South Alabama, Mobile, Alabama
  - University of Kansas Medical Center, Kansas City, Kansas
  - Children's Hospital Foundation Building, Louisville, Kentucky
  - Louisiana State University Health Sciences Center in New Orleans, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Detroit Medical Center (DMC), Detroit, Michigan
  - University Of Mississippi Medical Center, Jackson, Mississippi
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University Hospitals Case Medical Center-Case Western Reserve University (CWRU), Cleveland, Ohio
  - Regional Obstetrical Consultants, Chattanooga, Tennessee
  - The University of Texas Medical Branch (UTMB), Galveston, Texas
  - Texas Children's Hospital/Baylor College of Medicine, Houston, Texas
  - The University of Texas Health Science Center at Houston (UTHSC-H), Houston, Texas
  - Baylor Scott & White Health, Temple, Texas
  - University of Virginia School Of Medicine, Charlottesville, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Adalbertus Hospital, Gdansk, Pomeranian Voivodeship, Poland
- Sefako Makgatho Health Sciences University, Pretoria, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No